CLINICAL TRIAL: NCT03493529
Title: Microbiome and Endometrial Receptivity in Obese Infertile Women
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: IVI Bilbao (Other); IVI Barcelona (Other); Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: 1711-VLC-108-JB
Record Dates: First submitted 2018-03-08; First posted 2018-04-10 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Receptivity
Keywords: Endometrial microbiome; Obesity; Bacterial pathogens; Dysbiosis; Endometrial receptivity
MeSH Terms: conditions — Obesity; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Samples of saliva, feces and endometrial fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Weight: BMI: Between 18.50 and 29.99 kg/m2
- Obesity Clas I: BMI between 30 and 34.99 Kg/m2
- Obesity Clas II: BMI between 35 and 39.99 Kg/m2
- Obesity Clas III: BMI> 40 Kg/m2

SUMMARY:
The objective of this project is the identification and quantification of the main bacterial communities present in the endometrial microbiota in obese infertile patients, to assess if there is an alteration of their composition dependent on the body mass index, and if such alteration it could influence the reduction of endometrial receptivity, demonstrated in obese women. If obese patients have an altered digestive microbiota and, at the same time, a lower endometrial receptivity, the investigator want to assess whether such reduction in receptivity may depend on an alteration in the endometrial microbiota, which in non-obese infertile patients has been shown to negatively influence the reproductive results

DETAILED DESCRIPTION:
The main objective of our study is to compare the composition of the endometrial microbiota between patients with normal weight and patients with obesity.

A. Secondary Objectives/research questions

* To analyze the composition of the digestive microbiota through samples of saliva and feces in infertile patients with normal weight and obesity.
* To assess whether there is a relationship between the body mass index (normal weight, obesity Class I, Class II, Class III) and the main bacterial species detected in endometrial fluid samples from infertile patients.
* To evaluate the influence of the digestive microbiota on the composition of the endometrial microbiota according to the body mass index in infertile patients.
* To evaluate if there is an influence of the endometrial microbiota on the results of endometrial receptivity analyzed with the non-invasive Endometrial Receptivity Array test (niERA)

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients undergoing artificial cycle with HRT.
* Normal uterus confirmed by ultrasound (absence of uterine pathology such as submucosal or intramural myomas> 4 cm that deform cavity, endometrial polyps or Müllerian anomalies, or adnexal as communicating hydrosalpinx).
* Negative serological tests for HIV, HBV, HCV, RPR

Exclusion Criteria:

* Taking prescribed antibiotics or using IUDs or contraceptives 3 months prior to taking the sample. NOTE: Patients who have taken prophylactic antibiotics for ovarian puncture may be included at least 1 month before taking the sample.
* Age> 45 years
* Uncorrected uterine pathology, uncorrected hydrosalpinx
* Recurrent miscarriage (≥2 spontaneous abortions) or failure of implantation (transfer of 6 embryos in day 3 or 4 blastocysts in a cycle of IVF or donation of oocytes without gestation)
* Existence of serious or uncontrolled bacterial, fungal or viral infections that, in the opinion of the principal investigator, could interfere with the participation of the patient in the study or in the evaluation of the results of the study.
* Any disease or medical condition that is unstable or could endanger the patient's safety and compliance in the study.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients with normal weight (BMI: between 18.50 and 29.99) and obesity (Class I: BMI between 30 and 34.99 Kg / m2, Class II: BMI between 35 and 39.99 Kg / m2, Class III: BMI> 40 Kg / m2) subjected to Hormonal Replacement Therapy (HRT).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Microbiological analysis of endometrial fluid samples through massive sequencing | 14 months
  Identification and quantification of the main bacterial communities present in the endometrial microbiota of obese and normal-weight infertile patients through the analysis of the endometrial fluid.

SECONDARY OUTCOMES:
Microbiological analysis of saliva samples through massive sequencing. | 14 months
  Identification and quantification of the main bacterial communities present in the oral microbiota of obese and normal-weight infertile patients through the analysis of saliva samples.
Microbiological analysis of feces samples through massive sequencing. | 14 months
  Identification and quantification of the main bacterial communities present in the intestinal microbiota of obese and normal-weight infertile patients through the analysis of feces samples.
Analysis of endometrial receptivity using niERA | 13 months
  Analysis of the optimal implantation window through the study of the expression of 238 genes involved in receptivity using endometrial fluid samples.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE BELLVER PRADAS, MD, Principal Investigator — IVIRMA VALENCIA
Locations (1):
- Ivi Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No